CLINICAL TRIAL: NCT06149494
Title: A Trial in Participants With Chronic Obstructive Pulmonary Disease (COPD) to Evaluate the Impact of Vapendavir on the Development of Lower Respiratory Tract Symptoms Following Rhinovirus Challenge
Brief Title: RCT of Vapendavir in Patients With COPD and Human Rhinovirus/Enterovirus Upper Respiratory Infection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Altesa Biosciences, Inc. (Industry)
Collaborators: Virtus Respiratory Research (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ALT VPV-202
Record Dates: First submitted 2023-10-11; First posted 2023-11-29 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: COPD Exacerbation Acute; COPD With Acute Lower Respiratory Infection; Rhinovirus; Virus Diseases; Virus Infection, RNA; Enterovirus; Enterovirus Infections; Rhinovirus Infection; Infection Viral; Respiratory Complication; Respiratory Disease; Respiratory Tract Infections; Respiratory Tract Diseases; Respiratory Viral Infection; Upper Resp Tract Infection; Upper Respiratory Tract Infections; Upper Respiratory Disease; Upper Respiratory Disorder; Upper Respiratory Disease, Acute; Upper Respiratory Infection Viral; Infections, Respiratory; Infections; Copd; Viral Infection; Emphysema or COPD; Lower Respiratory Disease; Lower Respiratory Disorder; Lower Respiratory Tract and Lung Infections; Pulmonary Disease; Pulmonary Disease, Chronic Obstructive; Respiratory Disease Chronic; Lung Diseases; Lung Disease Chronic; Obstructive Pulmonary Disease; Chronic Lower Respiratory Diseases; Chronic Respiratory Disease
Keywords: Randomized; Double-blind; Phase 2; Placebo-Controlled; Clinical study; Clinical trial; Randomization; Interventional
MeSH Terms: conditions — Virus Diseases; RNA Virus Infections; Enterovirus Infections; Respiration Disorders; Respiratory Tract Infections; Respiratory Tract Diseases; Common Cold; Infections; Pulmonary Disease, Chronic Obstructive; Emphysema; Lung Diseases; Lung Diseases, Obstructive

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Vapendavir Cohort (Experimental): VPV will be dispensed by the study team on Day 0 at the clinical study visit at the study site. Participants will be given enough VPV for the 7-day treatment phase, (eg. Days 2 to 8). Treatment is twice daily, am and pm, 12 h apart ± 2 h. VPV micronized free base tablets (250 mg each) will be given orally beginning with a 1,000 mg loading dose (4 tablets) as soon as symptoms are present or the subject answers "yes" to "do you think you have a cold today" followed by 500 mg (2 tablets) either on the same day (eg day 2) or the next day. Treatment will therefore be for a total of 7 days consisting of an initial 1,000 mg dose (4-tablets) followed by thirteen 500mg doses (2-tablets). Treatment may occur within the home, on non-clinical study days.
  Interventions: Drug: Vapendavir
- Placebo Cohort (Placebo Comparator): Placebo will be dispensed by the study team on Day 0 at the clinical visit at the study site. Participants will be given enough Placebo for the 7-day treatment phase, (eg. Days 2 to 8). Treatment is twice daily, am and pm, 12 h apart ± 2 h. Placebo tablets will be matched to the active treatment and will be administered orally for 7 days as follows: 4 tablets for the initial dose as soon as symptoms are present or the subject answers "yes" to "do you think you have a cold today" on the first day of dosing (eg. Day 2), and 2 tablets, either on the same day (eg Day 2) or the next day. Treatment will therefore be for a total of 7 days (consisting of an initial 4-tablet dose followed by thirteen 2-tablet doses). Treatment may occur within the home, on non-clinical study days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Vapendavir — Participants randomized to the experimental cohort will be administered Vapendavir.
  Arms: Vapendavir Cohort
Drug: Placebo — Participants randomized to the placebo cohort will be administered placebo.
  Arms: Placebo Cohort

SUMMARY:
Vapendavir (VPV) is a drug being developed to treat human rhinovirus (RV) infection, one virus responsible for the common cold. Vapendavir prevents the virus from entering cells and making more infectious copies of itself. A study is being planned to investigate VPV in patients with chronic obstructive pulmonary disease (COPD, a lung disease making it difficult to breathe) who develop a rhinoviral infection; however, VPV has not been approved for use in treating any indication (disease) by the FDA or any other global regulatory agency. Therefore, VPV is considered investigational, and the study doctor is conducting this investigational research study. Safety will be monitored throughout the entire study.

DETAILED DESCRIPTION:
Study Drug Indication:

* Treatment of HRV infections in patients with COPD

Study Rationale:

An effective, easily administered therapy for RV infection would have the potential to reduce the serious health effects in vulnerable populations, such as those with COPD. Treatment of RV infection could reduce the severity and frequency of acute COPD exacerbations, preserve pulmonary function, prevent secondary bacterial infections, and mitigate the need for costly medical interventions, including inhaled agents, steroids, antibacterial drugs, emergency treatment, hospitalization, and mechanical ventilation. Thus, early treatment of acute COPD exacerbations related to RV infection could potentially improve both the quality of life and longevity of COPD patients.

Altesa BioSciences, Inc. is developing drugs to treat RV and other respiratory virus infections. VPV has been shown to inhibit RV in vitro and in human clinical trials. Furthermore, VPV has been administered to more than 650 study participants and has been well-tolerated. Based on its potential to prevent severe respiratory complications, Altesa BioSciences, Inc is continuing the development of this drug for the treatment of RV infection.

Study Dose justification:

* In patients with asthma, vapendavir doses of 264 mg bid and 528 mg bid were utilized and demonstrated reduced viral load and was well tolerated.
* A PK study established the pharmacokinetics of a free based micronized tablet in achieving adequate plasma levels after a single dose in fed adults.

Study Treatment Duration:

* 7 days

End of Study:

* Up to 63 days, including the screening and follow-up periods.

Study Centers:

* There will be 1 study centre, ICRRU within Imperial College Healthcare NHS site at St Mary's Hospital London, United Kingdom.

Study Treatment:

* 1:1 randomization to Vapendavir 500mg bid or placebo

Study Procedures:

* Screening period (Pregnancy test for females, Lung function tests (FEV1, FVC, PEF), Height and Weight/BMI Calculation, Physical Examination, Vital Signs, Medical and Surgical history, Blood sample, COPD assessment test)
* Baseline visit to clinic (Pregnancy test for females, Physical examination, Safety assessments, Vital Signs, Concomitant medication assessment, Nasal lavage/nasosorption, Chest X-Ray, ECG, Blood for hematology, biochemistry and liver function tests, Induced Sputum, Lung Function Tests (FEV1, FVC, PEF))
* Clinical Visit Day 1 (Randomization to treatment, Dispense Medication, Physical Examination, Safety Assessments, Vital Signs, Concomitant medication assessment, Nasal lavage/nasosorption, Chest X-Ray, ECG, Blood for hematology, biochemistry and liver function tests, Induced Sputum, Lung Function Tests (FEV1, FVC, PEF), Intranasal RV-A16 challenge)
* Treatment Commencement-Clinical Visit Days 1-28 (Physical Exam, Safety Assessments, Vital Signs, Concomitant Medication and food assessments, Diaries and eCRF completion, Treatment twice daily (If required), Drug Compliance, Nasal Lavage/nasosorption, Blood serum for biomarkers, Blood for hematology and biochemistry, Blood for PK, Pregnancy test for females, Lung Function Tests (FEV1, FVC, PEF))
* Treatment Commencement-Clinical Visit Day 42 (Physical Examination, Safety Assessments, Vital Signs, Concomitant medication and food assessments, Diaries and eCRF completion, Nasal lavage/nasosorption, Blood serum for biomarkers, blood for hematology, biochemistry and liver function tests, Blood sample taken to assess RV-A16 sero-positivity, Pregnancy test for females, Lung Function Tests (FEV1, FVC, PEF))
* Early Termination Visit (Physical Examination, Safety Assessments, Vital Signs, Concomitant medication and food assessments, Diaries and eCRF completion, Nasal lavage/nasosorption, Blood Serum for Biomarkers, Blood for hematology and biochemistry, Blood for PK, Sputum
* Unscheduled Visit (Physical Examination, Safety Assessments, Vital Signs, Concomitant medication and food assessments, Diaries and eCRF completion, Drug complicance, Lung function tests (FEV1, FVC, PEPF), Blood or PK-morning (or sampling))
* Study drug administered as soon as possible after onset of symptoms and documentation of HRV infection, but no greater than 48 hours after symptom onset.

Study Sample Size:

• 50 participants randomization will be 1:1 VPV : placebo. Participants will undergo 7 days of twice daily treatment. Treatment will commence after symptom onset or when the participant determines they have a clinical cold.

Statistical Methods:

* Efficacy Analysis: All participants infected and treated will comprise the infected and evaluable population and be included in the efficacy analysis (primary, secondary, exploratory endpoints). Subjects inoculated but not successfully infected will not be included in this analysis.
* Safety Analysis: All participants that have undergone any treatment with VPV or placebo will comprise the safety population and will be included in the safety analysis. Subjects that are inoculated, treated but not successfully infected will be included in this population.
* Inoculated & Followed-Up Population: Participants that are inoculated, but that do not fit the criteria to undergo treatment or become pregnant will be followed up until Day 42 ± 2. This group will be composed of both uninfected and successfully infected participants and follow up will be to obtain data on the RV challenge model, COPD related symptoms and also for safety reasons.
* Statistical Analysis Plan: A comprehensive Statistical Analysis Plan (SAP) will be finalized prior to reporting of the study results. The SAP may modify the plans outlined in the protocol; however, any major modifications of planned analyses will be reflected in a protocol amendment.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female age ≥40 years and ≤75 years at the time of signing the informed consent form.
2. If sexually active and/or of child-bearing potential (both females and males), must agree to use a highly effective forms of contraception ≥ 28 days prior to the first dose (females), during the study period (both males and females) and for 30 days (females) or 90 days (males) after the last dose. A woman is considered of childbearing potential (WOCBP), i.e. fertile, following menarche and until becoming post-menopausal unless permanently sterile. Permanent sterilisation methods include hysterectomy, bilateral salpingectomy and bilateral oophorectomy. A postmenopausal state is defined as no menses for 12 months without an alternative medical cause. A high follicle stimulating hormone (FSH) level in the postmenopausal range may be used to confirm a postmenopausal state in women not using hormonal contraception or hormonal replacement therapy. However, in the absence of 12 months of amenorrhea, a single FSH measurement is insufficient. Highly effective contraception is defined as methods that can achieve a failure rate of less than 1% per year when used consistently and correctly.

   Males (including those with a vasectomy): agree to use a condom and if a female partner of childbearing potential, use of at least one other contraceptive method; males must also agree not to donate sperm within 90 days after the last dose).

   WOCBP participants must use at least one highly effective contraceptive method.

   Birth control methods which may be considered as highly effective:
   * Combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation

     * oral
     * intravaginal
     * transdermal
   * progestogen-only hormonal contraception associated with inhibition of ovulation

     * oral
     * injectable
     * implantable
   * intrauterine device (IUD)
   * intrauterine hormone-releasing system ( IUS)
   * bilateral tubal occlusion
   * vasectomised partner
3. Confirmed diagnosis of Global Initiative for Chronic Obstructive Pulmonary Disease (GOLD) stage II COPD as defined by % predicted Forced expiratory volume in 1 second (FEV1) ≥50% and FEV1/Forced vital capacity (FVC) <70%.
4. History of acute exacerbations of COPD as defined by the participant answering "yes" to the question "do your COPD symptoms get noticeably worse when you catch a cold?"
5. If on maintenance therapy, be medically stable for at least 2 months prior to enrolment.
6. Clinically stable with no exacerbations within 2 months prior to enrolment.
7. Ability to understand and give informed consent.

Exclusion Criteria:

1. Participants with other causes of chronic airflow limitation:

   1. Including but not limited to: Asthma (mixed COPD and asthma is acceptable); cystic fibrosis (CF); bronchiolitis obliterans; and fibrosis such as tuberculosis (TB), idiopathic pulmonary fibrosis (IPF), or other major respiratory diagnosis (e.g., pneumonia, aspergillosis), etc.
   2. Non-CF bronchiectasis
2. Any disorder, for example, cardiovascular, gastrointestinal, hepatic, renal, neurological, musculoskeletal, infectious, endocrine, metabolic, haematological, psychiatric impairment that is not medically stable, or other major physical impairment that is not considered by the investigator medically stable/controlled.
3. Prescription or over-the-counter medications or herbal products that could be impacted by CYP3A4 and CYP 2C19 induction or inhibition and have serious complications for the participant within the treatment period without the ability to discontinue safely with a sufficient washout period before initiating VPV.
4. Patients on oral contraceptives or estrogen containing hormone replacement therapy.
5. Ingestion of grapefruit, pomegranate, star fruit and Seville oranges within 14 days prior to dosing. The juices and products containing these fruits should also be avoided.
6. History of clinically significant infection (respiratory or non-respiratory) requiring antibiotic or systemic steroids >10 mg/day within 30 days prior to planned RV challenge.
7. Pregnant, planning to become pregnant, testing positive for pregnancy at the screening visit test, or nursing females during and within 30 days of treatment.
8. Any cold symptom within the last 6 weeks such as sore throat, sneezing, rhinorrhoea, malaise, nasal obstruction or cough.
9. Presence (at screening) of serum rhinovirus 16 neutralising antibody titers at greater than or equal to one in four (≥1/4) dilution.
10. Active allergic rhinitis, active nasal disease such as nasal polyposis, chronic rhinosinusitis etc.
11. Active alcohol and/or drug misuse, at the discretion of the Investigator.
12. Use of any over the counter cold prophylaxis products including nasal sprays, C-vitamins, zinc or Echinacea within 1 month prior to the enrolment.
13. Participation in other clinical trial with medical investigational product within 30 days or 5 drug half-lives (whichever is longer) prior to enrolment.
14. Hypersensitivity/allergy to any of the active or placebo ingredients/ components.
15. Individuals with close contact to at risk patient group, including:

    * Infants (less than 6 months);
    * The extremely elderly or infirm;
    * Pregnant and/or breastfeeding women;
    * Patients with immunosuppression (e.g., human immunodeficiency virus (HIV), transplant recipients on anti-rejection medications, those undergoing chemo- or immuno-therapy).
    * Other factors that in the opinion of the investigator are considered a risk.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2023-11-20 (Actual); Primary Completion 2025-03-30 (Actual); Study Completion 2025-03-30 (Actual)

PRIMARY OUTCOMES:
Peak change from baseline | From Baseline Visit through Follow-Up Visit, up to 7 weeks
  • Evaluation of the peak total lower respiratory symptom score (LRSS) in participants administered with VPV relative to/versus (vs) placebo as determined by Mallia et al (Am J Respir Crit Care Med. 2011) from day of treatment commencement until Day 42. This is a measure of a number of lower respiratory symptoms in a 24 hour period that include: shortness of breath (scale 0-4; 0 = not breathless, 4 = breathless at rest) wheeze (0-4; 0 = no wheeze, 4 = wheeze at rest), cough (0-3; 0 = no cough, 3 = severe cough), sputum quantity (0-3; 0 = none, 3 = large volume , more than 100 ml) sputum quality (0-3; 0 = none, 3 = purulent, green in colour). The total lower respiratory symptom score is the sum of all the above measurements (minimum 0, maximum 17) recorded on each day. These values will be recorded via a study diary over a six week period (day 0-42). Peak value is the highest daily total value over the 6 week post-infection period.

SECONDARY OUTCOMES:
Peak COPD Specific Respiratory Symptoms | Day of treatment commencement to Day 42
  The Exacerbations of Chronic obstructive disease Tool-Respiratory Symptoms (EXACT-RS), out of 40 and EXACT-PRO, out of 51. Each questionnaire asks questions about severity of symptoms and impact on daily tasks (reach scored 0-3 or 0-4, 0=not at all, 3 or 4=extremely.
Peak Upper Respiratory Symptoms | Day of treatment commencement to Day 42
  Jackson Score as measured by Mallia et al (Am J Respir Crit Care Med. 2011). A modified Jackson score will be utilized which assesses the following eight upper respiratory symptoms daily: nasal congestion, runny nose, sneezing, cough, sore throat, general malaise, headache, chilliness (each scored 0-3 where 0 = none, 3 = severe). Minimum daily score= 0, maximum daily score= 24.
Peak Overall Symptom severity | Day of treatment commencement to Day 42
  * Patient global impression of severity (PGIS) The PGIS asks one question on disease severity and is scored from 0-3 (0=none, 3=severe)
  * Patient global impression of change (PGIC). The PGIC asks one question on how symptoms have changed from yesterday (-3 to +3 where -3= much worse, 0=no change and +3= much better).
Peak Virus Load as measured in RNA copies per mL | Day of treatment commencement to Day 42
  * Nasal lavage virus load
  * Sputum virus load
Peak Sputum Bacterial Load | Day of treatment commencement to Day 42
  * Total 16SrRNA as measured in DNA copies per mL
  * Moraxella catarrhalis as measured in DNA copies per mL
  * Streptococcus pneumoniae as measured in DNA copies per mL
  * Haemophilus influenzae as measured in DNA copies per mL
  * Bacterial load as measured in pfu per mL by NHS microbiology culture
Maximum Change in Forced Expiratory Volume in 1 Second (FEV1) | Day of treatment commencement to Day 42
  * FEV1 as measured in L/second
  * FEV1 as measured in % predicted from L/second
Maximum Change in Forced Vital Capacity | Day of treatment commencement to Day 42
  * Forced Vital Capacity (FVC) as measured in L
  * FVC as measured in % predicted from L
Maximum Change in FEV1/FVC | Day of treatment commencement to Day 42
  FEV1/FVC ratio in L

CONTACTS AND LOCATIONS:
Overall Officials: Onn Min Kon, MD, Principal Investigator — Imperial College Healthcare
Locations (1):
- St. Mary's Hospital - Imperial College Respiratory Research Unit (ICRRU), London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Sponsor website — https://www.altesabio.com/